CLINICAL TRIAL: NCT01488422
Title: Structural and Functional Mechanisms of Stress Reduction
Brief Title: Neural Correlates of Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AT006344
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Stress; Psychological Stress; Life Stress; Emotional Stress; Social Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Both groups will receive stress reduction materials. We expect both groups to achieve similar amounts of stress reduction, but to use different brain regions to do so.
  Interventions: Behavioral: Stress Reduction
- Group 2 (Active Comparator): Both groups will receive stress reduction materials. We expect both groups to achieve similar amounts of stress reduction, but to use different brain regions to do so.
  Interventions: Behavioral: Stress Reduction

INTERVENTIONS:
Behavioral: Stress Reduction — We are comparing 2 well-studied approaches to stress reduction. All participants will receive stress reduction instructions that have already been proven to effectively reduce stress. Our goal is to compare the neural mechanisms associated with both approaches.

SUMMARY:
This study will identify neural mechanisms associated with changes in emotion regulation following participation in stress reduction programs.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Right-handed
* Stressed

Exclusion Criteria:

* Lifetime history of schizophrenia or psychosis
* Psychiatric illness
* History of seizure or significant head trauma
* Use of psychotropic medications
* Metallic implants or devices contraindicating magnetic resonance imaging
* Claustrophobia
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in gray matter structure | 8 weeks
  Study participants will undergo an MRI scan before and after attending an 8-week stress reduction program.

SECONDARY OUTCOMES:
Emotion regulation | 8-weeks
  Study participants will do an emotion regulation task while they are in the MRI scanner. We will assess brain activity and skin conductance during the task. Changes in these measures will be assessed before and after enrollment in the stress reduction program

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sevinc G, Holzel BK, Greenberg J, Gard T, Brunsch V, Hashmi JA, Vangel M, Orr SP, Milad MR, Lazar SW. Strengthened Hippocampal Circuits Underlie Enhanced Retrieval of Extinguished Fear Memories Following Mindfulness Training. Biol Psychiatry. 2019 Nov 1;86(9):693-702. doi: 10.1016/j.biopsych.2019.05.017. Epub 2019 May 30. PMID 31303261